CLINICAL TRIAL: NCT00068055
Title: A Phase I/II Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of Intravenous Immunoglobulin G (OMR-IGG-AM) Containing High Anti-West Nile Virus Antibody Titers in Patients With, or at High Risk for Progression to West Nile Virus (WNV) Encephalitis and/or Myelitis
Brief Title: IVIG - West Nile Encephalitis: Safety and Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-107; CASG 210
Record Dates: First submitted 2003-09-04; First posted 2003-09-08 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2009-07

CONDITIONS: West Nile Virus
Keywords: West Nile Virus, encephalitis, myelitis, immunoglobulin G
MeSH Terms: conditions — Encephalitis; Myelitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): 60 subjects to receive Omr-IgG-am.
  Interventions: Drug: Omr-lgG-am
- 2 (Active Comparator): 20 subjects to receive Polygam® S/D (IVIG).
  Interventions: Drug: Polygam® S/D
- 3 (Placebo Comparator): 20 subjects to receive normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omr-lgG-am — Omr-IgG-am™ 5% is provided in 100 ml bottles (5.0 grams) as a sterile solution containing 5% protein, 10% maltose and water for injection. This product is licensed in Israel, but not in the US.
  Arms: 1
Drug: Polygam® S/D — Polygam® S/D is a solvent/detergent treated, sterile, freeze-dried preparation of highly purified immunoglobulin G (IgG) derived from large pools of human plasma. When reconstituted (5%) with the supplied diluent (sterile water for injection, USP) Polygam® S/D contains approximately 50mg of protein per ml (approximately 90% is gamma globulin); 3mg/ml human albumin, 22.5 mg/ml glycine, 20 mg/ml glucose, 2mlg/ml polyethylene glycol (PEG), 1 mcg/ml tri-nbutyl phosphate, 1 mcg/ml octoxynol 9, and 100 mcg/ml polysorbate 80.
  Arms: 2
Drug: Placebo — Normal Saline.
  Arms: 3

SUMMARY:
This study will look at the safety and effectiveness of an experimental medication containing antibodies (Omr-IgG-am™) in people with West Nile Virus (WNV) who already have brain and/or spinal cord inflammation or who are at high risk of developing these problems because they have weak immune systems. WNV can cause problems such as headaches, fever, muscle weakness, coma, and death. Study investigators believe people who are not able to fight infection well may be at risk for developing neurologic problems (having to do with the brain, spinal cord, nerves, and muscles) if they get WNV infection. Up to 110 subjects, 18 years or older, will participate for about 3 months and will receive either Omr-IgG-am™, Polygam® S/D, or placebo given through a small tube placed in a blood vessel in the arm. Hospitalization, up to 5 additional study visits, blood sample collection, MRI pictures of the brain and spinal cord, and neurological, muscle, and heart activity tests are also required.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether Omr-IgG-am™, an intravenous immunoglobulin (IVIg) containing antibodies specific for West Nile virus (WNV), is safe and well-tolerated in patients with suspected or laboratory diagnosed WNV disease. An initial estimation of efficacy will also be made. This Phase I/II study will enroll hospitalized adults with a presumptive diagnosis of West Nile encephalitis and/or myelitis or those with a positive laboratory test for diagnosis of WNV infection who are at high risk for progressing to severe neurologic disease based on age or immunosuppression. Patients will be randomized in blocks of five to receive either Omr-IgGam ™, Polygam® S/D (IVIG containing minimal anti-WNV antibodies) or normal saline in a ratio of 3:1:1. Patients and investigators will be blinded to treatment assignments. Patients will receive a single intravenous dose of study medication or one of two placebos. The study participants will receive 0.5 grams/kg of Omr-IgG-am™ or Polygam® S/D or a comparable volume of normal saline. All patients will be followed for safety, natural history endpoints, and efficacy. A subset of patients will have pharmacokinetic measurements of specific anti-WNV antibodies assessed following treatment. The primary endpoints are safety and tolerability following Omr-IgG-am™ administration. Secondary endpoints include pharmacokinetics of specific anti-WNV antibodies, mortality in confirmed WNV positive patients, and the combination of mortality and functional status at three months in both confirmed WNV-infected patients and all patients by intention to treat. This combined endpoint will be measured using four standardized measures of cognitive and functional status: the Barthel Index; the Modified Rankin Scale; the Glasgow Outcome Score; and the Modified Mini-Mental Status Examination. A comparison of outcomes will be made for the group receiving Omr-IgG-am™ versus those receiving either placebo, and between the two placebo groups. Other secondary endpoints include the proportion of patients in each group returning to pre-morbid baseline and each subject's improvement at 3 months as compared to that subject's worst (of any previous) evaluation. Natural history endpoints will also be assessed. They will include the duration of intensive care unit and hospital stay, development and persistence of WNV-specific IgG and IgM antibodies, combined functional score and mortality at 3 months between the group with encephalitis and/or myelitis at baseline versus the group with a positive WNV test only, outcomes in patients treated late in coma and correlation of outcome with time-to-treatment following symptom onset.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this clinical trial, all subjects (or legal representative) must provide written informed consent. Only patients meeting entry criteria will be enrolled. Eligible subjects must fall into one of two categories:

A. Hospitalized patients greater than or equal to 18 years of age with encephalitis and/or myelitis as defined below:

New neurologic abnormality:

* Asymmetric extremity weakness without sensory abnormality; or
* Other neurologic abnormality (including altered level of consciousness, dysarthria and dysphagia) plus fever (subjective or objective) within the previous 4 days AND

CSF examination within the previous 96 hours showing:

* Absence of organism on gram or fungal stain
* White blood cell count greater than or equal to 4 per cubic mm corrected for significant red blood cell contamination.
* Ratio of CSF: plasma glucose of greater than or equal to 40% (CSF glucose / plasma glucose greater than or equal to 0.4) Serum and CSF glucose levels should be obtained within 8 hours of each other for this calculation.

OR

B. Hospitalized patients, without encephalitis and/or myelitis as defined below, who meet the following criteria:

A positive IgM serology or PCR test for WNV in blood or cerebrospinal fluid, AND

Clinical illness compatible with WNV infection as described by occurrence of greater than or equal to 3 of the following findings during the preceding less than or equal to 10 days:

* Diarrhea
* Headache
* Fever > 38º C
* Nausea and/or vomiting
* Myalgias and/or arthralgias
* Nuchal rigidity
* Macular or papular rash
* New neurological abnormality AND

A risk factor for the development of WNV neurologic disease as defined by:

* Age greater than or equal to 40 years, or
* Age greater than or equal to 18 years plus immunosuppression, as defined by any of the following:

Hematologic malignancy; previous diagnosis of diabetes mellitus; chemotherapy within previous 4 weeks; stem cell transplant recipient or solid organ transplant recipient; taking immunosuppressive medications, including prednisone greater than or equal to 7.5 mg/day within the previous 4 weeks; history of human immunodeficiency virus (HIV) infection, congenital immunodeficiency syndrome (including common variable immunodeficiency)

Exclusion Criteria:

Unable to obtain valid informed consent History of intolerance (including anaphylaxis) to IVIg or related compounds Known history of IgA deficiency Known history of hypersensitivity to maltose

History of (or at time of study entry) hyperviscosity syndrome, such as but not limited to:

* Waldenstrom's macroglobulinemia
* Multiple myeloma
* Total white blood cell count > 80,000/cubic mm
* Hematocrit > 55%
* Platelet count > 700,000/cubic mm Meets criteria of Class III or IV of the New York Heart Association Classification for congestive heart failure patients Serum creatinine > 2.5 mg/dL or requires dialysis Alternate explanation (as determined by the investigator) for clinical findings (such as structural brain lesion, cerebrovascular accident, or other infectious disease, including confirmed infections with other flaviviruses) Pregnant or breastfeeding (negative serum or urine pregnancy test within previous 72 hours if woman is not postmenopausal or has not been surgically sterilized) Investigator's opinion that patient would be unable to adhere to protocol requirements Receipt of ribavirin, interferon alpha, intravenous immunoglobulin, or any investigational drug for treatment of WNV or hepatitis within 15 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2003-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety (including all causes of mortality) in the test IVIg (Omr-IgG-am™) group versus the 2 placebo groups, as defined by the total number of serious adverse events regardless of relatedness to study drug administration. | Duration of study.

SECONDARY OUTCOMES:
Pharmacokinetics of specific anti-WNV antibodies as measured by ELISA and PRNT methods. | Baseline (pre-dose) blood sample collected immediately prior to the beginning of the infusion. After the infusion, additional blood samples collected at 1 hr, 6 hr, 12 hr, 24 hr, 72 hr, and then at Day 5, Day 7, Day 14, Day 30, Day 60 and Day 90.
Proportion of patients returning to pre-morbid baseline at 3 months, between treated and untreated groups of patients with WNV infection, as assessed by two scoring systems the Barthel Index and the MRS. | At 3 months.
Improvement as compared to subject's own worst (of any earlier) evaluation, for each subject as defined by the combined results of the 4 neurological functional tests. | At 3 months.
Mortality alone among confirmed WNV patients. | At 3 months.
Combined morbidity and mortality in treatment versus placebo groups for all (including those without WNV infection) subjects by intention to treat analysis. | At 3 months.
Combined primary endpoint of mortality and morbidity among confirmed WNV patients as assessed by four scoring systems: the Barthel Index, the MRS, the GOS and the 3MS, in the experimental treatment group versus the control group. | At 3 months.

CONTACTS AND LOCATIONS:
Locations (69):
- United States (66):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Enloe Medical Center, Chico, California
  - Seton Medical Center, Daly City, California
  - City of Hope National Medical Center, Duarte, California
  - Kaiser Permanente South Bay Medical Center, Harbor City, California
  - University of Southern California, Los Angeles, California
  - University of California Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Santa Rosa Kaiser Medical, Santa Rosa, California
  - Exempla St. Joseph Hospital, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Infectious Disease Specialists, PC, Missoula, Montana
  - Central Nebraska Medical Clinic, Broken Bow, Nebraska
  - McCook Clinic, PC, McCook, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - VA Medical Center - Omaha, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Clara Maass Medical Center, Belleville, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Flushing Hospital Medical Center, Flushing, New York
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Dakota Clinic at Innovis, Fargo, North Dakota
  - MeritCare Hospital, Fargo, North Dakota
  - Trinity Health - Hospital, Minot, North Dakota
  - University Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson AFB, Ohio
  - Legacy Good Samaritan, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Infectious Disease Consultations - Rapid City, Rapid City, South Dakota
  - Avera Research Institute, Sioux Falls, South Dakota
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Medical Branch, Galveston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
  - Wilford Hall Medical Center, San Antonio, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba